CLINICAL TRIAL: NCT03594513
Title: Comparison Between Porcine Acellular Dermal Matrix (Mucoderm®) Versus Connective Tissue Graft in the Treatment of Multiple Adjacent Gingival Recessions Associated With Non-carious Cervical Lesion Partially Restored.
Brief Title: Mucoderm® Versus CTG in the Treatment of Multiple Gingival Recessions Associated With Non-carious Cervical Lesion.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Associate professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR
Record Dates: First submitted 2018-06-21; First posted 2018-07-20 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Gingival Recession; Tooth Abrasion
Keywords: Gingival Recession; Tooth Abrasion; Mucoderm
MeSH Terms: conditions — Gingival Recession; Tooth Abrasion | interventions — Drug Prescriptions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCAF+PR+CTG (Active Comparator): The partial restoration of the NCCL will be performed prior the surgeries and will be carried out with composite resin.The surgical procedure for root coverage will be carried out by means modified coronally advanced flap and will be performed by starting with oblique incisions in the interdental areas, which continued with the intrasulcular incision at the recession defects.Each surgical papilla will be dissected in a split-thickness and the envelope flap will be raised with a split-full-split thickness in the coronal-apical direction. Additionally, this group will receive the connective tissue graft harvested from the palate on the recessed area before the sutures.Then, the flap will be coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: MCAF; Procedure: PR; Procedure: CTG; Drug: Sodium dipyrone; Drug: chlorhexidine rinse
- MCAF+PR+XMD(Mucoderm®) (Experimental): The partial restoration of the NCCL will be performed prior the surgeries and will be carried out with composite resin.The surgical procedure for root coverage will be carried out by means modified coronally advanced flap and will be performed by starting with oblique incisions in the interdental areas, which continued with the intrasulcular incision at the recession defects.Each surgical papilla will be dissected in a split-thickness and the envelope flap will be raised with a split-full-split thickness in the coronal-apical direction. Additionally, this group will receive a porcine acellular dermal matrix on the recessed area before the sutures. Then, the flap will be coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: MCAF; Procedure: PR; Procedure: XMD(Mucoderm®); Drug: Sodium dipyrone; Drug: chlorhexidine rinse

INTERVENTIONS:
Procedure: MCAF — Periodontal surgical technique to treat gingival recessions.
  Other Names: Periodontal plastic surgery
Procedure: PR — Restorative procedure to treat tooth structure loss.
  Other Names: Composite resin restoration
Procedure: CTG — Autogenous graft harvested from palate placed in the surgical site.
  Other Names: Connective tissue graft
  Arms: MCAF+PR+CTG
Procedure: XMD(Mucoderm®) — Xenogenous graft placed in the surgical site.
  Other Names: Porcine acellular dermal matrix
  Arms: MCAF+PR+XMD(Mucoderm®)
Drug: Sodium dipyrone — All participants were instructed to take 500 mg sodium dipyrone just in case of pain.
  Other Names: Drug prescription
Drug: chlorhexidine rinse — All participants were instructed to perform 0.12% chlorhexidine rinse after the surgical procedures.
  Other Names: Drug prescription

SUMMARY:
The aim of the present study is to compare two different multidisciplinary protocols using two types of grafts, porcine acellular dermal matrix (Mucoderm®) versus connective tissue graft, both associated with modified coronally advanced flap, in the treatment of multiple adjacent gingival recessions associated with non-carious cervical lesion partially (NCCL) restored by composite resin.

DETAILED DESCRIPTION:
This is a prospective, parallel and controlled clinical trial assessing non-inferiority in root coverage and superiority in oral health-related quality of life. The population that will be evaluated in this is study will be enrolled at São Paulo State University (Unesp), Institute of Science and Technology, São José dos Campos.

Forty patients with multiple adjacent gingival recessions associated with non-carious cervical lesion will be enrolled and randomly allocated to one of the following groups:

* Test group (n=20): partial restoration of cervical lesion and modified coronally advanced flap for root coverage associated with porcine acellular dermal matrix (MCAF+PR+XMD)
* Control group (n=20): partial restoration of cervical lesion and modified coronally advanced flap associated with connective tissue graft (MCAF+PR+CTG).

The restorative treatment of non-carious cervical lesion will be performed one week prior the surgical procedures and will be conducted as follows. After local anesthesia, rubber dam isolation will be placed, and a coronal bevel will be performed at the incisal margin of the NCCL to reduce the step of lesions and to allow a correct and harmonious emergence profile of the restoration. Afterward, acid etching with 37% phosphoric acid will be performed and washed for 30 seconds with water-air-jet. The lesion will be dried with sterile cotton pellets to prevent dehydration, and the adhesive will be applied according to the manufacturer's instructions (Single Bond Universal, 3M ESPE). The adhesive will be light cured for 20 seconds, and the restoration will be made with resin composite (Filtek Z350 XT, 3M ESPE). The apical margin of the restoration will be determined to be 1 mm apical to the estimated position of the cementoenamel junction(CEJ) in order to rebuild only the anatomical part of the crown destroyed by the NCCL and 1 mm of the root surface, once the apical portion of the root surface will be covered by gingival tissue after periodontal surgery. After rubber dam removal, the restoration will be finished with ultrafine-grained burs, and 48 hours after the restoration procedure, polishing will be completed with diamond paste and felt discs.

All surgeries will be performed by the same expert periodontist (MPS). The surgical procedure for root coverage will be carried out according to Zucchelli's technique (Zucchelli et al., 2000). In brief description, following local anesthesia, oblique submarginal incisions in the interdental areas, which continued with the intrasulcular incision at the recession defects, will be carried out keeping a blade 15c (Swann-Morton® - Sheffield, England) mounted on No. 3 scalpel handle parallel to the long axis of the teeth to dissect in a split-thickness manner the surgical papilla. Each surgical papilla will be dislocated with respect to the anatomic papilla by the oblique submarginal interdental incisions. The envelope flap will be raised with a split-full-split thickness in the coronal-apical direction: gingival tissue apical to the root exposures will be raised in a full-thickness manner to provide that portion of the flap critical for root coverage with more thickness and the most apical portion of the flap will be elevated in a split-thickness manner to facilitate the coronal displacement of the flap. The portion of the root exposure with loss of clinical attachment will be instrumented with the use of curets. The remaining tissue of the anatomic interdental papilla will be de-epithelialized to create connective tissue beds to which the surgical papilla will be sutured through sling sutures to coronally cover 2 mm above the CEJ after the placement of the grafts. For the test group (MCAF+PR+XMD), a porcine acellular dermal matrix (Mucoderm®, Botiss, Berlin, Germany) will be trimmed with a scalpel in appropriate shape and size to cover the root surfaces and underlying bone. Lastly, for the control group (MCAF + PR + CTG), a connective tissue graft will be harvested from the palate according to Bruno's technique (Bruno JF, 1994).

After the surgery, the participants will be requested to take 500 mg of sodium dipyrone every 8 hours for 3 days in case of pain and to avoid brushing and flossing in the treated area for a period of 2 weeks. During this period, plaque control will be achieved using 0.12% chlorhexidine solution twice a day. The sutures will be removed after 10 days, and all of the patients will be recalled for prophylaxis and reinforcement of motivation and instruction for atraumatic toothbrushing during the study period.

Clinical, esthetics, and comfort of patients parameters will be assessed at 45 days, 2, 3 and 6 months after the surgical procedure.

Quantitative data will be recorded as mean ± standard deviation (SD), and normality will be tested using Shapiro-Wilk tests. The probing depth (PD), relative gingival recession (RGR), clinical attachment level (CAL), keratinized tissue thickness (KTT), keratinized tissue width (KTW), and dentin hypersensitivity (DH) values will be examined by two-way repeated measures ANOVA to evaluate the differences within and between groups, followed by a Tukey test for multiple comparisons when the Shapiro-Wilk p value was ≥ 0.05. Those presenting Shapiro-Wilk p values < 0.05 will be analyzed using a Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Patient's esthetics and discomfort measures using, respectively, visual analog scale (VAS) and postoperative diary (Tonetti et al. 2018) will be analyzed by T-tests. The frequency of complete root coverage will be compared using χ2 tests. Intergroup root coverage esthetic score (RES) comparisons will be performed with a T-test. A significance level of 0.05 will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting three or more Miller class I or II multiple adjacent gingival recessions (recession depth ≥ 2,5 mm) in incisors, canines or premolars associated with non-carious cervical lesion;
* teeth included in the study should present pulp vitality;
* patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤ 20%;
* patients older than 18 years old;
* probing depth ˂ 3 mm in the included teeth;
* patients who agreed to participate and signed an informed consent form.

Exclusion Criteria:

* patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure
* patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure
* smokers or pregnant women
* patients who underwent periodontal surgery in the area of interest;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of defect coverage | 6 months
  Percentage mean (%) of root surface covered by the surgical treatment, measured through a periodontal probe.

SECONDARY OUTCOMES:
Modified root coverage esthetic score | 6 months
  The Modified Root Coverage Esthetic Scale (MRES; Santamaria et al. 2014) will be performed by two blinded and independent examiners at the 6-month post-operative assessment. This score evaluates six variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, gingival color, and restoration/cervical lesion color.
Dentine hypersensitivity | 6 months
  Evaluation of root sensitivity with the air blow test and measurement with a visual analog scale (VAS).
Patient recovery | 14 days
  Evaluation of postsurgery sequelae, pain, and discomfort, oral function and interference with daily activities through postoperative diary previously described (Tonetti et al. 2018).
Patient-centred esthetic evaluation | 6 months
  Esthetic evaluation performed by the patient through a visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP
Locations (1):
- São Paulo State University, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zucchelli G, De Sanctis M. Treatment of multiple recession-type defects in patients with esthetic demands. J Periodontol. 2000 Sep;71(9):1506-14. doi: 10.1902/jop.2000.71.9.1506. PMID 11022782
- [Background] Tonetti MS, Cortellini P, Pellegrini G, Nieri M, Bonaccini D, Allegri M, Bouchard P, Cairo F, Conforti G, Fourmousis I, Graziani F, Guerrero A, Halben J, Malet J, Rasperini G, Topoll H, Wachtel H, Wallkamm B, Zabalegui I, Zuhr O. Xenogenic collagen matrix or autologous connective tissue graft as adjunct to coronally advanced flaps for coverage of multiple adjacent gingival recession: Randomized trial assessing non-inferiority in root coverage and superiority in oral health-related quality of life. J Clin Periodontol. 2018 Jan;45(1):78-88. doi: 10.1111/jcpe.12834. Epub 2017 Nov 21. PMID 29087001
- [Background] Bruno JF. Connective tissue graft technique assuring wide root coverage. Int J Periodontics Restorative Dent. 1994 Apr;14(2):126-37. PMID 7928129
- [Background] Silveira CA, Mathias IF, da Silva Neves FL, Castro Dos Santos NC, Araujo CF, Neves Jardini MA, Bresciani E, Santamaria MP. Connective Tissue Graft and Crown-Resin Composite Restoration for the Treatment of Gingival Recession Associated with Noncarious Cervical Lesions: Case Series. Int J Periodontics Restorative Dent. 2017 Jul/Aug;37(4):601-607. doi: 10.11607/prd.3044. PMID 28609509